CLINICAL TRIAL: NCT06806605
Title: Full-3D Computer-Assisted Workflow for the Diagnosis and Correction of Deformities? Dentofacial
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: FULL-3D OS
Record Dates: First submitted 2024-11-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Dentofacial Deformities
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- T0 Initial 3D study: T0: the patient has not yet started orthodontic-surgical treatment and is carrying out the initial documentation collection;
  Interventions: Other: 3d analisys
- T1 Preoperative 3D study: T1: the patient one month before surgery who collects the preoperative documentation;
  Interventions: Other: 3d analisys
- T2 Final 3D study: T2: the patient has completed the orthodontic-surgical treatment and performs the collection of the final documentation. It is carried out within 12 months of the intervention.
  Interventions: Other: 3d analisys

INTERVENTIONS:
Other: 3d analisys — To analyze the orthodontic-surgical set-up carried out as part of the normal care pathway of patients operated since January 2015 and who completed treatment on May 30, 2020 in the Orthodontic First patient.

SUMMARY:
"Dentofacial deformity refers to deviations from the norm of facial proportions and tooth ratios of such magnitude as to represent a disability." [1] These conditions afflicted two aspects of the patient's health: the first related to the functions performed by the stomatognathic apparatus (mastication, swallowing, phonation, etc...), the second related to the morphology of the face, which--by virtue of the severe disharmony of its parts--did not fully realize its function as an organ of relationships, leading the patient to high levels of psychological distress.

The nature of the dentofacial deformities was mainly related to skeletal discrepancies between the maxillae, such that the malocclusion could not be resolved by orthodontic treatment alone. The resolution of these conditions required a perfect synergy between orthodontic therapy (aimed at dental alignment of the individual arches) and surgical therapy (aimed at morphological harmonization of the face and obtaining the correct occlusion).

DETAILED DESCRIPTION:
**Orthognathic Surgery**

Orthognathic surgery allows the repositioning of the jaws in all three spatial planes. This procedure is indicated for patients with:

* Class 3 malocclusion, caused by maxillary retrusion, mandibular prognathism, or a combination of the two;
* Class 2 malocclusion, due to mandibular retrusion, with a normally conformed, protruded, or retruded maxilla and/or with excessive verticality;
* Class 1 malocclusion, characterized by consensual bimaxillary retrusion (a condition that may be seen in complex medical issues, such as in OSAS patients);
* Facial asymmetries caused by overgrowth on one side or facial torsion;
* Other malocclusions not correctable with orthodontic treatment alone, such as transversal or dento-alveolar deficits;
* Sequelae from facial trauma.

Orthognathic surgery has progressed rapidly since the 1950s when surgical techniques for treating most malocclusions that could not be resolved through orthodontics alone were first developed.

Subsequent technological advances have simplified the diagnosis of dentofacial deformities in three dimensions: Multislice CT (MSCT), Cone Beam CT (CBCT), Magnetic Resonance Imaging (MRI), stereophotogrammetry, dental arch scanning, software that allows surgical planning and outcome prediction, intraoperative navigation, and CAD-CAM technology. The conventional approach to orthognathic surgery (Orthodontic-first) consists of three phases: pre-surgical orthodontic treatment, the surgical phase, and post-surgical occlusion stabilization (post-surgical orthodontic treatment).

**Orthognathic Surgery and Technology: From 2D Study to 3D** To diagnose dentofacial deformities, the investigators have utilized 3D digital records created through dedicated software or devices. Real data and digital information are combined to simulate the surgical procedure.

**3D Cephalometry** Cephalometry is the method used to analyze the geometry of facial structures. Historically, this method was based on 2D radiology. The use of CT allowed the application of the same geometric criteria to 3D reconstructions of the skull and face. Studies assessing its accuracy showed that this method is comparable to standard 2D cephalometry for known measurements, but it adds a significant amount of new information, particularly regarding the rotational and translational aspects of the jaws and individual teeth.

**3D Surgical Planning** It is now possible to plan surgery using computer-assisted digital methods. The surgical plan can be transferred accurately to the patient through CAD-CAM-manufactured devices. The planning process can simulate both orthodontic and/or surgical treatment.

At the University of Bologna, the investigators have extensive experience with intraoperative navigation guided by 3D virtual simulation, combining navigation and virtual 3D surgery. they also have expertise in producing individualized CAD-CAM synthesis devices. It has been previously demonstrated that virtual orthodontic planning is as reliable as traditional methods using plaster models in orthodontic-only patients.

In fact, incorporating digital orthodontic planning into the orthodontic/surgical workflow is of great importance for the following reasons:

1. Initial treatment prediction to better guide therapeutic choices;
2. Improved communication between orthodontists and surgeons;
3. Enhanced communication with patients, providing an accurate prediction of the treatment plan from the beginning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dentoskeletal dysmorphia.
* Patients undergoing orthognathic surgery.
* Patients between 18 and 60 years of age at the time of orthognathic surgery.
* Obtaining informed consent.Inclusion criteria
* Patients with dentoskeletal dysmorphia.
* Patients undergoing orthognathic surgery.
* Patients between 18 and 60 years of age at the time of orthognathic surgery.
* Obtaining informed consent.

Exclusion Criteria:

* Patients who have undergone other facial surgeries during the treatment period.
* Patients who have not followed the data collection phases foreseen in the 3D Study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients operated since January 2015 and who completed the "T2" follow-up by May 30, 2020, at the Maxillofacial Surgery Department (AOU di Bologna), who followed the normal care pathway provided for cases of dentoskeletal dysmorphosis, which consisted of:
  T0: Initial 3D study (before the start of orthodontic treatment) T1: Preoperative 3D study (1 month after surgery) T2: Final 3D study (at the end of post-operative orthodontic treatment with the appliance removed)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
primary outcome | 18 months
  The primary outcome are :
  analyze the surgical orthodontic set-up at time T0 (pre-treatment phase) in relation to the decompensation orthodontics actually performed and the surgery actually planned at time T1 (pre-operative phase).

SECONDARY OUTCOMES:
secondary outcome | 18 months
  evaluate the accuracy of the surgical orthodontic set-ups performed at time T0 and T1 in relation to the results obtained at the end of the treatment in the patient at time T2 (patient who has completed the surgical orthodontic treatment).

OTHER OUTCOMES:
pre-specified outcomes | 18 months
  * "T0": the patient has not yet started orthodontic-surgical treatment and performs the initial documentation collection;
  * "T1": the patient one month before surgery who performs the collection of the pre-operative documentation;
  * Surgical intervention;
  * "T2": the patient has completed orthodontic-surgical treatment and who performs the collection of the final documentation. It is performed within 12 months of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Marchetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided